CLINICAL TRIAL: NCT04092816
Title: The Fathers and Mothers Invested in Lives of Their Youth (FAMILY) Study: A Pilot Intervention for Families Affected by Parental Cancer
Brief Title: Fathers and Mothers Invested in Lives of Their Youth (FAMILY) Study: A Pilot Intervention
Acronym: FAMILY
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped prematurely due to difficulty meeting accrual and retention goals, exacerbated by the COVID-19 pandemic.
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LCCC1920; 5K07CA218167-02 (NIH)
Record Dates: First submitted 2019-09-04; First posted 2019-09-17 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Metastatic Breast Cancer; Parenting
Keywords: Parenting
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: 10 patient and co-parent dyads (20 participants in total) will participate in the pilot study to evaluate the feasibility and acceptability of the FAMILY intervention. Preliminary effects of the intervention will also be examined.
Masking Description: Because this is a pilot study, all participant dyads will receive the same intervention and no blinding will take place.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FAMILY (Experimental): Patient-co-parent dyads will participate in the FAMILY intervention in-person.
  Interventions: Behavioral: FAMILY Intervention

INTERVENTIONS:
Behavioral: FAMILY Intervention — The FAMILY intervention involves 2-3 study visits with a specially-trained intervention facilitator. Study visits are manualized and complemented by patient education materials.

SUMMARY:
This is a single-arm pilot study to evaluate the feasibility and acceptability of a novel psychosocial intervention to improve psychosocial outcomes for parents with advanced cancer and their co-parents. In this single-center study, we will recruit ten mothers with metastatic breast cancer and their co-parents as dyads (N=20) to participate in the Fathers and Mothers Invested in the Lives of their Youth (FAMILY) intervention. Patient and co-parent dyads will participate in 2-3 study visits with an intervention facilitator and a post-intervention feedback interview. Participants will also complete baseline and follow-up study surveys. The final products of this study will be the FAMILY intervention manual and training materials, and fidelity assessments.

DETAILED DESCRIPTION:
Cancer is the leading disease-specific cause of early parental death in the United States and having dependent children worsens suffering for parents with advanced cancer and their families. The FAMILY intervention consists of manualized visits with a trained intervention facilitator and psychoeducation materials to help parents cope with cancer-related parenting concerns. The purpose of the intervention is to improve parenting concerns, emotional well-being, and end-of-life (EOL) preparation among participants. This study will evaluate whether a psychosocial intervention to reduce psychological distress and improve EOL preparation for mothers with metastatic breast cancer and their co-parents can be acceptable, feasible, and relevant to the target patient population.

This study is needed in order to generate critical data to: (1) refine the intervention in preparation for a pilot efficacy randomized controlled trial (RCT); and to generate preliminary data demonstrating the feasibility and acceptability of core intervention components. The preliminary data will support future grant applications for a full-scale efficacy RCT.

ELIGIBILITY:
Inclusion Criteria for patients:

* Be a woman with metastatic (stage IV) breast cancer who has either: (1) estrogen (ER), progesterone (PR), or HER2 receptor-negative cancer and disease progression beyond first line of therapy, or (2) ER, PR, or HER2 -positive cancer and disease progression beyond two lines of therapy;
* A mother of at least one dependent child, defined as a child <18 years of age who lives at least half-time in the home;
* Be at least 18 years of age;
* Adequate stamina to complete at least two study visits
* Able to provide informed consent
* Able to complete all study measures and visits in English;
* Be willing to participate in study visits at the North Carolina Cancer Hospital (NCCH) if they live >75 miles away from NCCH
* Have an identified co-parent who is eligible and willing to participate in the study.

Inclusion Criteria for Co-parents:

* Be an adult man or woman who is both a partners or spouse of the patient and who would serve as the child(ren)'s primary caregiver if the patient were to become unavailable;
* Able to provide informed consent;
* Able to complete all study measures and visits in English;
* Stated willingness to comply with all study procedures; and
* Be at least 18 years of age.

Exclusion Criteria for patients and co-parents:

* Unable to participate in study visits due to illiteracy, inability to speak English or other causes.
* Live more than 75-miles away from the North Carolina Cancer Hospital (NCCH) and unable to attend study visits at NCCH (participants who live more than 75-miles away and can attend study visits at NCCH remain eligible for participation).
* Unwilling to be audio-recorded during facilitated study visits and feedback interview.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zev M Nakamura, MD, Principal Investigator — University of North Carolina
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 10/30/2019 through 01/25/2022 at one cancer center in North Carolina.
Pre-assignment Details: A total of 15 subjects (8 patients and 7 co-parents) consented and were found eligible for the study.
Groups:
- Patients: Subjects who are diagnosed with cancer.
- Co-parents: Subjects who are spouses of patients with cancer.
Period: Overall Study
Arm/Group | Patients | Co-parents
Started | 5 | 5
Completed | 4 | 3
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Population: Eight patients and 7 co-parents consented.
Groups:
- Patient: Subjects who are diagnosed with cancer.
- Co-parent: Subjects who are spouses of patients with cancer.
- Total: Total of all reporting groups
Arm/Group | Patient | Co-parent | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.75 (8.65) | 45.67 (10.21) | 42.86 (9.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 0 | 8
  Male | 0 | 7 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of the Intervention
Description: Acceptability of the intervention was defined as the number of participants who completed the study intervention. Participants' experience was assessed qualitatively, using post-intervention interviews.
Time Frame: 42 Days
Population: The number of total participants who started the intervention and completed post-intervention semi-structured interview.
Measure: Count of Participants; unit: Participants
Arm/Group | FAMILY
Number analyzed (Participants) | 10
Participants
  The patient and co-parent started the study. | 10
  The patient and co-parent completed a post-intervention interview. | 7

2. Primary Outcome: Acceptability of the Intervention Measured by the Study Visit Assessment Form
Description: The acceptability of the intervention was assessed through participants' satisfaction with the program. The Lyon Satisfaction questionnaire consists of 5-point Likert-type items assessing positive (six items) and negative (seven items) emotional reactions to the study visit. Responses were summed and reported for each subscale with higher scores meaning higher emotional reactions, and worse reactions. Positive subscale: 6-30 and negative subscale: 7-35.
Time Frame: 7 Days
Population: 10 Subjects completed the study visit assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAMILY
Number analyzed (Participants) | 10
score on a scale
  Positive emotions | 26.6 (5.3)
  Negative emotions | 11.7 (2.8)

3. Primary Outcome: Feasibility of Study Procedures
Description: Feasibility of study procedures were assessed how likely patient-co-parent dyads are to join the study through tracking the number of eligible dyads who participate in the study.
Time Frame: 14 Days
Population: The number of participants (patient and co-parent) who started the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients | Co-parents
Number analyzed (Participants) | 5 | 5
Participants
  Started | 5 | 5
  Completed | 4 | 3

4. Primary Outcome: Feasibility of Recruitment
Description: Assess how likely patient-co-parent dyads are to join the study by tracking the number of eligible dyads who participate in the study.
Time Frame: Baseline
Population: All 18 participants/co-parents were approached by the study team.
Measure: Count of Participants; unit: Participants
Groups:
- Patients: Subjects with a cancer diagnosis.
- Co-parents: Subjects who are spouse of a patient with cancer diagnosis.
Arm/Group | Patients | Co-parents
Number analyzed (Participants) | 9 | 9
Participants
  Eligible | 9 | 9
  Consented | 8 | 7

5. Secondary Outcome: Feasibility of Completion
Description: Feasibility of Completion was evaluated by tracking the number of dyads that complete the study visits and study assessments. Numbers reflect from Baseline through 42 days given a flexible duration of intervention.
Time Frame: Up to 42 Days
Population: The number of participants (patient and co-parent) consented and completed study visits.
Measure: Count of Participants; unit: Participants
Groups:
- Patiens: Subjects who are diagnosed with cancer.
Arm/Group | Patiens | Co-parents
Number analyzed (Participants) | 8 | 7
Participants
  Enrolled | 8 | 7
  Baseline | 6 | 5
  7 days | 5 | 5
  14 days | 4 | 3
  28 days | 2 | 2
  42 days | 0 | 0

6. Secondary Outcome: Emotional Well-being Measured by the Functional Assessment of Chronic Illness Therapy - Palliative Care (FACIT-Pal Care) Subscale
Description: Assess the change in patient's emotional well-being through the FACIT-Pal Care; a 6-item self-report assessment of emotional well-being that is widely used in palliative care research. Score range is 0-24, higher scores indicate better emotional well-being.
Time Frame: Baseline, 7 Days, 14 Days, 28 Days, 42 Days
Population: Baseline, patient participants only
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FAMILY
Number analyzed (Participants) | 5
units on a scale
  Baseline | 16.4 (4.3)
  7 days | 18.0 (4.5)
  14 days: number analyzed (Participants) | 3
  14 days | 13.7 (1.2)
  28 days: number analyzed (Participants) | 2
  28 days | 20.5 (2.1)
  42 days: number analyzed (Participants) | 0

7. Secondary Outcome: Anxiety and Depression Symptoms Measured by the Hospital Anxiety and Depression Scale (HADS)
Description: Assess the change in patient and co-parent's depression and anxiety symptom severity. The HADS consists of two 7-item subscales assessing depression and anxiety symptoms separately. Score range for each subscale is 0-21, higher scores indicate greater symptoms.
Time Frame: Baseline, 7 Days, 14 Days, 28 Days, 42 Days
Population: Numbers analyzed reflect participants at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAMILY
Number analyzed (Participants) | 10
score on a scale
  Baseline Anxiety | 8.6 (2.8)
  Baseline Depression | 5.1 (3.8)
  7 Days Anxiety | 8.1 (2.4)
  7 Days Depression | 5.7 (4.3)
  14 Days Anxiety: number analyzed (Participants) | 7
  14 Days Anxiety | 9.0 (1.7)
  14 Days Depression: number analyzed (Participants) | 7
  14 Days Depression | 6.0 (4.3)
  28 Days Anxiety: number analyzed (Participants) | 4
  28 Days Anxiety | 9.3 (2.2)
  28 Days Depression: number analyzed (Participants) | 4
  28 Days Depression | 3.3 (2.2)
  42 Days Anxiety: number analyzed (Participants) | 0
  42 Days Depression: number analyzed (Participants) | 0

8. Secondary Outcome: Parenting Concerns Measured by the Parenting Concerns Questionnaire-Advanced Disease (PCQ-AD)
Description: Assess the change in patient and co-parent's parenting concerns severity. The PCQ-AD is an investigator-adapted measure of parenting concerns measured on a 4-point scale. Total score range for the PCQ-AD is 0-3 with higher scores indicating greater distress.
Time Frame: Baseline, 7 Days, 14 Days, 28 Days, 42 Days
Population: Number analyzed reflects the number of participants at each time point contributing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAMILY
Number analyzed (Participants) | 10
score on a scale
  Baseline | 1.8 (0.6)
  7 Days | 1.5 (0.7)
  14 Days: number analyzed (Participants) | 7
  14 Days | 1.5 (0.6)
  28 Days: number analyzed (Participants) | 4
  28 Days | 1.1 (0.4)
  42 Days: number analyzed (Participants) | 0

9. Secondary Outcome: The Change in Patient and Co-parent's Illness-related Communication
Description: The change in patient and co-parent's illness-related communication was measured by the Couples Illness Communication Scale (CICS).
  The CICS is a brief self-report measure of illness-related couple communication. The CICS consists of 4 items measured on a 5-point Likert-type scale. Total Score Range: 4-20, Higher is better.
Time Frame: Baseline, 7 Days, 14 Days, 28 Days, 42 Days
Population: Numbers reflect participants at each time point given flexible duration of intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAMILY
Number analyzed (Participants) | 10
score on a scale
  Baseline | 12.5 (3.0)
  7 Days | 14.1 (2.2)
  14 Days: number analyzed (Participants) | 7
  14 Days | 13.6 (4.5)
  28 Days: number analyzed (Participants) | 4
  28 Days | 14.3 (4.4)
  42 Days: number analyzed (Participants) | 0

10. Secondary Outcome: Patient's Health-related Quality of Life
Description: Patient Health-related Quality of Life was assessed change in the patient's health-related quality of life measured by the Functional Assessment of Chronic Illness Therapy - Palliative Care (FACIT-Pal).
  The FACIT-Pal is a 46-item self-administered assessment of general HRQOL in cancer patients. It is graded on a 4-point scale and higher scores indicate better quality of life. Total Score Range: 0-184
  Assess change in the patient's health-related quality of life measured by the FACIT-Pal; the FACIT-Pal is a 46-item self-administered assessment of general HRQOL in cancer patients. It is graded on a 4-point scale and higher scores indicate better quality of life.
  The numbers analyzed reflect all individuals who contributed data at each time point.
Time Frame: Baseline, 7 Days, 14 Days, 28 Days, 42 Days
Population: Only patient participants completed the measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAMILY
Number analyzed (Participants) | 5
score on a scale
  Baseline | 122.8 (36.1)
  7 Days | 122.8 (44.4)
  14 Days: number analyzed (Participants) | 4
  14 Days | 138.7 (24.1)
  28 Days: number analyzed (Participants) | 2
  28 Days | 162.5 (0.7)
  42 Days: number analyzed (Participants) | 0

11. Secondary Outcome: Patient and Co-parent's Cancer-related Family Communication
Description: Patient and Co-Parent's Cancer-related Family Communication was assessed changes in the patient and co-parent's scores for a nine-item investigator-developed measure.
  The measure assesses participants' confidence and preparation to engage in communication about the impact of parental cancer on children. For the first 8 items, the score range is on a 4-point scale (1 to 4). The last item is graded on a 3-point scale (1 to 3). For all 9 items, higher is better. Due to the small sample size, each individual score item was reported.
Time Frame: Baseline, 7 Days, 14 Days, 28 Days, 42 Days
Population: Numbers analyzed reflect all participants who contributed data at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAMILY
Number analyzed (Participants) | 10
score on a scale
  Baseline - comfort talking with children | 2.8 (1.0)
  Baseline - comfort talking with partner | 3.7 (0.5)
  Baseline - comfort talking about children's future needs | 3.4 (1.0)
  Baseline - prepared to talk with children | 2.7 (0.9)
  Baseline - prepared to talk with partner | 3.5 (0.7)
  Baseline - prepared to talk about children's future needs | 3.5 (0.7)
  Baseline - understand partner | 1.4 (0.7)
  Baseline - spending time with children | 3.6 (1.4)
  Baseline - prior conversations with children | 1.9 (1.0)
  7 Days - comfort talking with children | 2.6 (0.8)
  7 Days - comfort talking with partner | 3.2 (0.4)
  7 Days - comfort talking about children's future needs | 3.5 (0.5)
  7 Days - prepared to talk with children | 2.5 (1.0)
  7 Days - prepared to talk with partner | 3.3 (0.5)
  7 Days - prepared to talk about children's future needs | 3.3 (0.5)
  7 Days - understand partner | 1.4 (0.5)
  7 Days - spending time with children | 4.6 (0.7)
  7 Days - prior conversations with children | 2.0 (0.9)
  14 Days - comfort talking with children: number analyzed (Participants) | 7
  14 Days - comfort talking with children | 3.0 (1.0)
  14 Days - comfort talking with partner: number analyzed (Participants) | 7
  14 Days - comfort talking with partner | 3.0 (0.6)
  14 Days - comfort talking about children's future needs: number analyzed (Participants) | 7
  14 Days - comfort talking about children's future needs | 3.0 (0.6)
  14 Days - prepared to talk with children: number analyzed (Participants) | 7
  14 Days - prepared to talk with children | 3.0 (0.6)
  14 Days - prepared to talk with partner: number analyzed (Participants) | 7
  14 Days - prepared to talk with partner | 3.3 (0.5)
  14 Days - prepared to talk about children's future needs: number analyzed (Participants) | 7
  14 Days - prepared to talk about children's future needs | 3.3 (0.5)
  14 Days - understand partner: number analyzed (Participants) | 7
  14 Days - understand partner | 1.1 (0.4)
  14 Days - spending time with children: number analyzed (Participants) | 7
  14 Days - spending time with children | 4.1 (0.7)
  14 Days - prior conversations with children: number analyzed (Participants) | 7
  14 Days - prior conversations with children | 2.1 (0.9)
  28 Days - comfort talking with children: number analyzed (Participants) | 4
  28 Days - comfort talking with children | 3.0 (0.8)
  28 Days - comfort talking with partner: number analyzed (Participants) | 4
  28 Days - comfort talking with partner | 3.3 (0.5)
  28 Days - comfort talking about children's future needs: number analyzed (Participants) | 4
  28 Days - comfort talking about children's future needs | 3.3 (0.5)
  28 Days - prepared to talk with children: number analyzed (Participants) | 4
  28 Days - prepared to talk with children | 3.0 (0.8)
  28 Days - prepared to talk with partner: number analyzed (Participants) | 4
  28 Days - prepared to talk with partner | 3.0 (1.0)
  28 Days - prepared to talk about children's future needs: number analyzed (Participants) | 4
  28 Days - prepared to talk about children's future needs | 3.0 (1.0)
  28 Days - understand partner: number analyzed (Participants) | 4
  28 Days - understand partner | 1.5 (1.0)
  28 Days - spending time with children: number analyzed (Participants) | 4
  28 Days - spending time with children | 4.5 (0.6)
  28 Days - prior conversations with children: number analyzed (Participants) | 4
  28 Days - prior conversations with children | 2.0 (1.2)
  42 Days - comfort talking with children: number analyzed (Participants) | 0
  42 Days - comfort talking with partner: number analyzed (Participants) | 0
  42 Days - comfort talking about children's future needs: number analyzed (Participants) | 0
  42 Days - prepared to talk with children: number analyzed (Participants) | 0
  42 Days - prepared to talk with partner: number analyzed (Participants) | 0
  42 Days - prepared to talk about children's future needs: number analyzed (Participants) | 0
  42 Days - understand partner: number analyzed (Participants) | 0
  42 Days - spending time with children: number analyzed (Participants) | 0
  42 Days - prior conversations with children: number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Not available. The protocol does not require adverse event assessment.
Description: The protocol does not require adverse event assessment. Adverse Event Data was not collected.
Arm/Group | FAMILY
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Early termination due to COVID-19 pandemic limiting research enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/16/NCT04092816/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT04092816/ICF_001.pdf